CLINICAL TRIAL: NCT07190378
Title: Predictive Factors of Steroid-Induced Diabetes and the Role of Continuous Glucose Monitoring in the Diagnosis and Metabolic Control of the Disease
Brief Title: Predictive Factors and Monitoring Strategies in Steroid-Induced Diabetes
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Jedrasek, Principal Investigator, Medical University of Warsaw
Other Study IDs: KB/90/2025
Record Dates: First submitted 2025-07-28; First posted 2025-09-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Steroid-Induced Diabetes; Diabete Type 2; Steroid Induced Hyperglycemia
Keywords: Steroid-induced diabetes; Steroid-induced hyperglycaemia; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with no prior history of diabetes initiating steroid therapy: Adult patient without history of diabetes, who are initiating steroid therapy will be enrolled in the study

SUMMARY:
Glucocorticoids are widely used in the management of autoimmune, inflammatory and neoplastic conditions. However, they are associated with significant metabolic effects, including steroid-induced diabetes (SID). SID is typically diagnosed using general criteria for type 2 diabetes, which may be inadequate due to the unique glycemic profile often seen in SID, where postprandial hyperglycemia predominates. This research aims to explore the diagnostic value of CGM during steroid therapy and identify risk factors for SID This is a prospective observational study (n=250) enrolling adults initiating glucocorticoid therapy. Participants will undergo 14-day continuous glucose monitoring (CGM) to assess predictive factors and glycemic profile.

DETAILED DESCRIPTION:
Approximately 250 patients hospitalised at Warsaw University Hospital will be enrolled. Baseline data collection includes medical history, anthropometry, HbA1c, and basic biochemical tests. CGM sensors will be applied. The glycemic profile will be monitored for 14 days using the CGM system. If time spent above 140 mg/dL exceeds 10%, capillary glucose testing will be used to confirm diabetes based on established clinical guidelines

ELIGIBILITY:
Inclusion criteria:

* Adults (≥18 years of age)
* No prior diagnosis of diabetes
* Planned initiation of oral and/or intravenous glucocorticoid therapy for non-substitutive indications
* Informed consent

Exclusion criteria:

* Age <18 years
* History of diabetes or use of antidiabetic medications
* GC therapy within the past 6 months
* Replacement therapy for primary or secondary adrenal insufficiency, pituitary insufficiency, Nelson's syndrome, or congenital adrenal hyperplasia
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with no prior history of diabetes initiating steroid therapy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2028-06-05 (Estimated); Study Completion 2028-06-19 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of diabetes | From enrollment to the end of the observation at 2 weeks
  diagnosis of steroid-induced diabetes based on fasting blood glucose 2 times above 126 mg/dl and/or HbA1c>6.5% and/or blood glucose above 200 mg/dl

SECONDARY OUTCOMES:
Glycemic Target | From enrollment to the end of the observation at 2 weeks
  Assessment of Time in range (70-180 mg/dl)
Time above 140 mg/dL for ≥10% of the day | From enrollment to the end of the observation at 2 weeks
  More than 10% of the day spend in range of glucose levels above 140 mg/dl is associated with significantly increased risk of diabetes
Hypoglycaemia Episodes | From enrollment to the end of the observation at 2 weeks
  Assessment of Time below range (<70 mg/dl) through Continuous Glucose Monitoring System
Glycemic profile | From enrollment to the end of the observation at 2 weeks
  Assessment of glycemic profile through CGM sensor: Glucose monitoring index

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Czupryniak, prof. dr hab. n. med., Study Director — Department of Diabetology and Internal Medicine, Medical University of Warsaw, Warsaw, Poland
Locations (1):
- Department of Diabetology and Internal Medicine, Medical University of Warsaw, Warsaw, Poland, Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No